CLINICAL TRIAL: NCT05425888
Title: Functional and Proprioceptive Status in Patients With Hemophilic Ankle Arthropathy. A Case-control Study
Brief Title: Functional and Proprioceptive Status in Patients With Hemophilic Ankle Arthropathy
Status: Completed | Type: Observational
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Collaborators: Real Fundación Victoria Eugenia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, Principal Investigator, University of Oviedo
Other Study IDs: He-AnkleCon
Record Dates: First submitted 2022-06-10; First posted 2022-06-21 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Haemophilia
Keywords: Hemophilic arthropathy; Ankle; Joint pain; Functionality; Range of motion; Proprioception
MeSH Terms: conditions — Hemophilia A; Arthralgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemophilia group: Group of adult patients with hemophilia, diagnosed with bilateral hemophilic ankle arthropathy
  Interventions: Other: Hemophilia group
- Control group: Group of healthy subjects with sociodemographic characteristics similar to patients with hemophilia, diagnosed with bilateral hemophilic ankle arthropathy.
  Interventions: Other: Hemophilia group

INTERVENTIONS:
Other: Hemophilia group — Evaluation of the study variables: dorsal flexion; dorsiflexion strength; tibialis anterior muscle activation; biomechanical analysis of gait and balance; and functionality.

SUMMARY:
Introduction: Hemophilic ankle arthropathy is manifested by functional degenerative alterations (muscle strength deficit, mobility and proprioception), intra-articular and chronic pain.

Design: Case-control study. Objective: To observe the differences between patients with hemophilic ankle arthropathy and their healthy peers, regarding dorsiflexion, dorsiflexion strength, biomechanical analysis of gait and balance, and functionality.

Patients: 10 patients with hemophilic ankle arthropathy and 12 healthy subjects without ankle joint damage.

Measurement instruments and study variables: dorsiflexion (range of motion), dorsiflexion strength (dynamometry), biomechanical analysis of gait and balance (RS SCAN® model platform), and functionality (2 Minute Walk Test).

Expected results: Analyze the main differences and their relationship based on the clinical and independent variables of patients with hemophilia, compared to their healthy peers.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A and B.
* Over 18 years.
* With medical diagnosis of ankle arthropathy.
* With clinical evaluation by Hemophilia Joint Health Score.
* In prophylactic treatment or on demand with FVIII / FIX concentrates for coagulation.
* No previous hemarthrosis of the ankles in the 3 months prior to evaluation.

Exclusion Criteria:

* Patients with inhibitors (antibodies against FVIII or FIX).
* Patients with neurological or cognitive disorders that prevent the understanding of questionnaires and physical tests.
* Failure to sign the informed consent document

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with hemophilic ankle arthropathy older than 18 years (group of cases). Healthy subjects without ankle joint damage, of the same age range (control groups).
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Assess the dorsal flexion with numerical scale of range of motion | Screening visit
  Measurement with Leg Motion system. Subjects will stand with the big toe on the starting line and the knee touching a metal stick. The metal rod will move away from the foot up to the maximum ankle dorsiflexion allowed, without taking the heel off the ground and with knee contact on the rod. Three measurements will be made for each ankle and the mean value will be used for data analysis. All measurements will be made with the patient barefoot.
Assess the dorsiflexion strength with dynamometry | Screening visit
  The maximal isometric strength of the ankle flexor muscles will be tested. Both extremities will be evaluated with a manual dynamometer (model Lafayette Manual Muscle Tester 01165). The examiner will hold the dynamometer on the sole of the foot while the subject exerts maximal force against it. The unit of measurement of this measurement instrument is the Newton per square centimeter (N/cm2), where the higher the score, the greater the muscle force.

SECONDARY OUTCOMES:
Assess the biomechanical analysis of gait and balance with pressure platform | Screening visit
  It will be evaluated using an Rs Scan® pressure platform and FootScan® pressure measurement system. This scientific version biomechanical examination device measures plantar pressure using an X-Y array of resistive pressure sensitive sensors that are scanned sequentially. The system records pressure data when the subject is standing or walking on the platform. Measurements will be made with the basic 0.5m platform with 4,096 sensors with resistive technology and 300Hz data acquisition frequency. The biomechanics of walking will be analyzed with the analysis of the probes and the static balance in a time of 30 seconds
Assess the functionality with pressure platform | Screening visit
  The 2-Minute Walking Test will be used. The functional capacity to exercise, in clinical practice, will be evaluated by means of a modified version, used in populations with pathologies with special characteristics, of the 6-minute version. It will be carried out in a closed corridor, with a length of 30 m delimited between cones. Before the test, participants must rest for at least 10 minutes. Subsequently, they will be instructed to complete the circuit by walking around the cones as fast as possible, but without running, for 2 minutes. They will be allowed to use walking aids, slow down or stop to rest if necessary. The distance covered at the end of the 2 minutes will be recorded by the evaluator. This instrument has shown excellent test-retest reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — University of Oviedo
Locations (1):
- Universidad Católica San Antonio, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided